CLINICAL TRIAL: NCT02333552
Title: A Cohort Study of Frailty Status Transition and Its Impact to Quality of Life in Outpatient Elderly
Brief Title: Frailty Status and Quality of Life in Elderly
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Siti Setiati, Prof. Siti Setiati, MD, PhD, SpPD-KGer, MEpid, Indonesia University
Other Study IDs: INA-FRAGILE00
Record Dates: First submitted 2015-01-02; First posted 2015-01-07 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Frailty; Quality of Life
Keywords: Frailty; Pre-frailty; Fit; Robust; Elderly; Sociodemography status; Functional status; Cognitive status; Nutrition status; Comorbidity; Mortality; Depression status
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Frailty is a dynamic process from fit (robust) and pre-frail elderly. There is no previous study that determine the risk factors from fit to pre-frailty and pre-frailty to frailty in Indonesian elderly.

This study was aimed to define the risk factors of frailty transitional status and its correlation with quality of life in Indonesian elderly outpatients.

DETAILED DESCRIPTION:
Frailty is an age-associated, biological syndrome characterized by decreased biological reserves, due to dysregulation of several physiological systems, which puts an individual at risk when facing minor stressors, and is associated with poor outcomes (ie, disability, death, and hospitalization).

Frailty identifies a high-risk subgroup and off ers characteristics of great clinical importance: a higher reversibility at early stages than disability, and a higher predictive value than chronic disease for adverse outcomes at older ages. It is also the most common condition leading to death in community-dwelling older people.

However, there is current consensus that physical frailty is potentially reversible. It is hence useful to objectively detect frailty among frail elderly persons, as frailty indices serve a useful purpose for risk stratification, predicting need for institutional care and planning of services needed.

To date, there is no study or information about frailty status in Indonesia elderly. This study was aimed to define the risk factors of frailty transitional status and its correlation with quality of life in Indonesian elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly aged >= 60 years old
2. Fit (robust) or pre-frailty;
3. Capable to understand and carry-out the instruction.

Exclusion Criteria:

1. Unwilling to join the study;
2. Abbreviated Mental Test (AMT) score < 8;
3. Geriatric Depression Scale (GDS) score >= 10;
4. Body mass index (BMI) <18,5 Kg/m2;
5. Malnutrition (according to Mini Nutritional Assessment/MNA);
6. Liver cirrhosis, severe liver dysfunction, or serum ALT levels >3 times upper normal limit;
7. Acute illness during inclusion period, eg. pneumonia, pain due to acute arthritis (visual analog scale >6/10), stroke attack, crisis hypertension;
8. Severe cardiac dysfunction: acute decompensated heart failure and/or chronic heart failure functional class III or IV (New York Heart Association classification);
9. Severe pulmonary dysfunction: acute exacerbation of chronic obstructive lung disease stage III or IV (GOLD classification), and/or PaO2 levels < 60 mmHg.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fit or pre-frail elderly aged >= 60 years old who came to Comprehensive Geriatric Clinics, Cipto Mangunkusumo General Hospital, Jakarta, during March 2013-April 2014.
Sampling Method: Non-Probability Sample
Enrollment: 269 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in frailty status at 24 months | Baseline and at 24 months
  Frailty status is divided into Fit (robust), Pre-frail, and Frailty.

SECONDARY OUTCOMES:
Change from baseline in mortality at 24 months | at 24 months
  Mortality: number of subjects died after 24 months observation.
Change from baseline in morbidities at 24 months | Baseline and at 24 months
  Morbidities: number of diseases in subjects (using Charlson Comorbidity Index)

CONTACTS AND LOCATIONS:
Overall Officials: Siti Setiati, Prof, MD, Principal Investigator — Division of Geriatrics, Department of Internal Medicine, Universitas Indonesia-Cipto Mangunkusumo General Hospital, Jakarta; Purwita Laksmi, MD, Study Chair — Division of Geriatrics, Department of Internal Medicine, Universitas Indonesia-Cipto Mangunkusumo General Hospital, Jakarta; Rahmi Istanti, SKM, MARS, Study Chair — Division of Geriatrics, Department of Internal Medicine, Universitas Indonesia-Cipto Mangunkusumo General Hospital, Jakarta

REFERENCES:
- [Background] Lee JS, Auyeung TW, Leung J, Kwok T, Woo J. Transitions in frailty states among community-living older adults and their associated factors. J Am Med Dir Assoc. 2014 Apr;15(4):281-6. doi: 10.1016/j.jamda.2013.12.002. Epub 2014 Feb 16. PMID 24534517
- [Background] Laksmi PW. Frailty syndrome: an emerging geriatric syndrome calling for its potential intervention. Acta Med Indones. 2014 Jul;46(3):173-4. No abstract available. PMID 25348178